CLINICAL TRIAL: NCT01371227
Title: A Phase 1 of JNS002 (Doxorubicin HCl Liposome Injection) in Combination With Bortezomib for Japanese Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of JNS002 (Doxorubicin Hydrochloride Liposome Injection) in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018085; JNS002-JPN-03 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-05-26; First posted 2011-06-10 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Relapsed or refractory multiple myeloma; JNS002; Bortezomib
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JNS002 (Experimental): JNS002 30 mg/m2 by intravenous infusion at a rate of = 1 mg/minute on Day 4 of each 21-day cycle.
  Interventions: Drug: JNS002

INTERVENTIONS:
Drug: JNS002 — 30 mg/m2 by intravenous infusion at a rate of = 1 mg/minute on Day 4 of each 21-day cycle.

SUMMARY:
The purpose of this study is to evaluate tolerability of the combination therapy of JNS002 and bortezomib in Japanese bortezomib-naive patients with multiple myeloma who have ever received at least 1 line of chemotherapy.

DETAILED DESCRIPTION:
This is a non-randomized (study drug is intentionally assigned to the patient), single-arm (one group of patients receiving the same treatment), open-label (all people involved know the identity of the intervention) study to evaluate tolerability of the combination therapy of JNS002 and bortezomib in 3 to 6 patients with multiple myeloma whose disease has either progressed after at least 1 line of prior therapy or was refractory to initial treatment. Initially, 3 patients will be enrolled and the incidence of dose limiting toxicity (DLT) will be determined at the end of Cycle 1 to evaluate the study doses against the maximum tolerated dose (MTD). If the incidence is =2/3, additional 3 patients will be enrolled to define the MTD. Safety endpoints include adverse events, laboratory tests (hematology, blood biochemistry, and urinalysis), electrocardiogram (ECG), LVEF, chest X-ray, vital signs (body temperature, pulse rate, and blood pressure), and body weight. Efficacy evaluation will be performed in terms of antitumor effect, according to criteria for assessment of antitumor effect similar to the European Group for Blood and Marrow Transplantation (EBMT) criteria. Bortezomib 1.3 mg/m2 by rapid (bolus) intravenous (IV) administration will be given on Days 1, 4, 8, and 11 of each 21-day cycle. In addition, JNS002 30 mg/m2 by IV infusion will be given at a rate of = 1 mg/minute on Day 4 of every 21-day cycle after bortezomib. Treatment will continue for a total of 6 cycles of therapy (126 days).

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed diagnosis of multiple myeloma with evaluable disease parameters (1.Presence of M-protein in the serum and/or urine, 2.Increased plasma cells in the bone marrow or biopsy-proven plasmacytoma, 3.Presence of related organ tissue impairment)
* Patients with progression of disease after an initial response (complete, partial, or minimal response based on the EBMT criteria) to at least 1 line of therapy. Progression of disease before responding to an initial line of therapy with a non-anthracycline containing regimen that included (at a minimum) an alkylating agent or high-dose corticosteroids. Rituximab alone or experimental agents alone were not to be considered a line of therapy
* Patients with progressive disease as defined by one of the following: i) > 25% increase in M-protein, ii) Development of new or worsening lytic bone lesions, iii) Development of new or worsening plasmacytoma, iv) Development of new or worsening hypercalcemia (> 11.5 mg/dL or 2.8 mmol/L corrected) that is not attributable to any other cause
* Patients with measurable secretory disease defined as either: i) Serum monoclonal protein > 1 g/dL, ii) Urine monoclonal (light chain) protein > 200 mg/24 hours
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1. ECOG performance status score 2 due to pain associated with bone disorder is eligible.

Exclusion Criteria:

* Patients with history of treatment with bortezomib
* Patients with progressive disease while receiving an anthracycline-containing regimen
* Patients with no change (NC) in disease status during initial therapy (patient must have had a response and then progression or progression while receiving initial therapy [primary refractory disease]
* Patients with non-secretory disease (i.e., no measurable paraprotein in serum or urine
* urine paraprotein level = 200 mg/24 hours)
* Patients with prior treatment with doxorubicin or other anthracycline at cumulative doses greater than 240 mg/m2 (calculated using doxorubicin equivalent doses: 1 mg doxorubicin = 1 mg JNS002 = 1.8 mg epirubicin = 0.3 mg mitoxantrone = 0.25 mg idarubicin)
* Patients with Grade 1 peripheral neuropathy with pain or Grade 2 or higher peripheral neuropathy, according to Common Terminology Criteria for Adverse Events (CTCAE)
* Patients with clinically significant heart disease, New York Heart Association (NYHA) Class II or higher heart failure
* Patients with viral hepatitis or chronic liver disease
* Patients with pulmonary fibrosis or interstitial pneumonitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | Up to 21 days

SECONDARY OUTCOMES:
Number of subjects who achieved a complete response or partial response | Up to 126 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (2):
- Japan (2):
  - Nagoya
  - Okayama

REFERENCES:
- [Derived] Kusumoto S, Sunami K, Inagaki M, Iida S. Phase I study of pegylated liposomal doxorubicin in combination with bortezomib for Japanese patients with relapsed or refractory multiple myeloma. Int J Hematol. 2015 Jun;101(6):578-84. doi: 10.1007/s12185-015-1773-5. Epub 2015 Mar 7. PMID 25749662
- See also: A Phase I Study of JNS002 (doxorubicin HCl liposome injection) in Combination with Bortezomib for Japanese Subjects with Relapsed or Refractory Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1111&filename=CR018085_CSR.pdf